CLINICAL TRIAL: NCT00004028
Title: PHASE I, OPEN LABEL, MULTICENTER DOSE ESCALATION STUDY OF GLIADEL IN PATIENTS WITH RECURRENT MALIGNANT GLIOMA
Brief Title: Carmustine in Treating Patients With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065129; NABTT-101-9601; JHOC-NABTT-101-9601; NCI-T96-0052H
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 1999-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult ependymoblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma; Neuroectodermal Tumors, Primitive; Gliosarcoma | interventions — Carmustine

INTERVENTIONS:
Drug: carmustine
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of carmustine in treating patients who are undergoing surgery for recurrent malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of polifeprosan 20 with carmustine implant (GLIADEL) in patients undergoing surgery for recurrent malignant glioma.

OUTLINE: This is a dose escalation study.

All patients undergo maximal tumor resection. At the time of surgery, groups of 6 patients receive up to 8 polifeprosan 20 wafers containing increasing doses of carmustine implanted into the resection cavity.

Patients with an intraoperative diagnosis other than glioblastoma multiforme or anaplastic astrocytoma do not receive wafer implantation, and are removed from study.

Patients are followed 3, 6, and 12 months after implantation.

PROJECTED ACCRUAL: A total of 52 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed recurrent malignant glioma for which surgery is indicated
* Unilateral, supratentorial, solitary lesion at least 1.0 cm in diameter on contrast-enhanced CT or MRI

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 8 weeks

Hematopoietic:

* WBC at least 3,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin, AST, ALT, and alkaline phosphatase less than 2.5 times normal

Renal:

* Creatinine less than 1.5 times normal
* BUN less than 2.5 times normal
* Protein no greater than 3 g/dL
* No gross hematuria

Other:

* No hypersensitivity to nitrosoureas
* Not pregnant
* Fertile patients must use effective contraception
* No concurrent life threatening disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent immunotherapy during first 8 weeks of study

Chemotherapy:

* At least 4 weeks since chemotherapy (6 weeks since nitrosoureas)
* No concurrent chemotherapy during first 8 weeks of study

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior definitive external-beam radiotherapy (i.e., at least 5,000 cGy) required
* No concurrent radiotherapy or brachytherapy during first 4 weeks of study

Surgery:

* Prior cytoreductive surgery for supratentorial brain tumor required
* Biopsy alone not sufficient

Other:

* No concurrent investigational therapy during first 8 weeks of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-09

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Olivi, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (9):
- United States (9):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Result] Olivi A, Grossman SA, Tatter S, Barker F, Judy K, Olsen J, Bruce J, Hilt D, Fisher J, Piantadosi S; New Approaches to Brain Tumor Therapy CNS Consortium. Dose escalation of carmustine in surgically implanted polymers in patients with recurrent malignant glioma: a New Approaches to Brain Tumor Therapy CNS Consortium trial. J Clin Oncol. 2003 May 1;21(9):1845-9. doi: 10.1200/JCO.2003.09.041. PMID 12721262